CLINICAL TRIAL: NCT03241706
Title: Effect of Liver Glycogen Content on Hypoglycemic Counterregulation
Brief Title: Liver Glycogen and Hypoglycemia in Humans
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jason Winnick (Other)
Responsible Party: Sponsor-Investigator, Jason Winnick, Assistant Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-7982
Record Dates: First submitted 2017-08-04; First posted 2017-08-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hypoglycemia; Iatrogenic
Keywords: hypoglycemia; type 1 diabetes; liver glucose metabolism
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Sodium Chloride; Somatostatin; Insulin; Glucagon; High Fructose Corn Syrup

STUDY DESIGN:
Who Masked: Participant
Masking Description: The subjects will not be informed which treatment they will receive for a given trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Controls-saline (Placebo Comparator): Each subject from Group 1 will undergo a metabolic study where saline is infused so as to not stimulate liver glucose uptake and glycogen deposition.
  Interventions: Drug: Saline; Drug: Somatostatin; Drug: Insulin; Drug: Glucagon; Drug: Dextrose solution
- Controls-high fructose (Active Comparator): A second group of control subjects will undergo a single metabolic study using a higher dose of fructose (6.5 mg/kg/min).
  Interventions: Drug: Low Fructose; Drug: Somatostatin; Drug: Insulin; Drug: Glucagon; Drug: Dextrose solution
- Controls-low fructose (Active Comparator): Each subject from Group 1 will undergo another metabolic study where fructose (1.3 mg/kg/min) is infused so as to stimulate liver glucose uptake and glycogen deposition.
  Interventions: Drug: Somatostatin; Drug: Insulin; Drug: Glucagon; Drug: Dextrose solution; Drug: High Fructose

INTERVENTIONS:
Drug: Low Fructose — IV fructose (1.3 mg/kg/min)
  Arms: Controls-high fructose
Drug: Saline — Saline given as a comparison to fructose.
  Arms: Controls-saline
Drug: Somatostatin — IV infusion of somatostatin (60 ng/kg/min)
  Other Names: SRIF
Drug: Insulin — IV infusion of insulin between 20-60 mU/m2/min.
Drug: Glucagon — IV glucagon (0.65 ng/kg/min).
Drug: Dextrose solution — IV dextrose to clamp the plasma glucose at the desired level.
  Other Names: d20
Drug: High Fructose — IV-fructose (6.5 mg/kg/min)
  Arms: Controls-low fructose

SUMMARY:
The purpose of this research study is to learn more about how sugar levels in the liver affect the ability of people both with and without type 1 diabetes. People with type 1 diabetes do not make their own insulin, and are therefore required to give themselves injections of insulin in order to keep their blood sugar under control. However, very often people with type 1 diabetes give themselves too much insulin and this causes their blood sugar to become very low, which can have a negative impact on their health. When the blood sugar becomes low, healthy people secrete hormones such as glucagon and epinephrine (i.e., adrenaline), which restore the blood sugar levels to normal by increasing liver glucose production into the blood. However, in people with type 1 diabetes, the ability to release glucagon and epinephrine is impaired and this reduces the amount of sugar the liver is able to release.

People with type 1 diabetes also have unusually low stores of sugar in their livers. It has been shown in animal studies that when the amount of sugar stored in the liver is increased, it increases the release of glucagon and epinephrine during insulin-induced hypoglycemia. In turn, this increase in hormone release boosts liver sugar production. However, it is not known if increased liver sugar content can influence these responses in people with and without type 1 diabetes. In addition, when people with type 1 diabetes do experience an episode of low blood sugar, it impairs their responses to low blood sugar the next day. It is also unknown whether this reduction in low blood sugar responses is caused by low liver sugar levels.

The investigators want to learn more about how liver sugar levels affect the ability to respond to low blood sugar.

DETAILED DESCRIPTION:
There is universal agreement that iatrogenic hypoglycemia is the single most prominent barrier to the safe, effective management of blood sugar in people with type 1 diabetes (T1D). The typical patient with T1D is required to "count" the number of carbohydrates they consume, estimate their own insulin doses and deliver this insulin subcutaneously to manage their own glycemic level. With these multiple degrees of freedom, it is not surprising that people with T1D frequently over-insulinize, thereby putting themselves at increased risk of developing hypoglycemia and its associated comorbidities.

As the glycemic level falls in people who are generally healthy (i.e., non-T1D), the first response is an abatement of insulin secretion. This reduction is then followed by an increase in the release of the counterregulatory hormones glucagon and epinephrine as glycemia continues to fall. Collectively, this hormonal milieu causes an increase in liver glycogen mobilization and gluconeogenesis such that hepatic glucose production (HGP) increases, thereby preventing serious hypoglycemia from occurring. However, people with T1D are unable to reduce their own insulin levels (due to subcutaneous insulin delivery) and often have a diminished capacity to secrete both glucagon and epinephrine during insulin-induced hypoglycemia. Predictably, the HGP response to hypoglycemia in people with T1D is a fraction of that seen in non-T1D controls, thereby increasing the depth and duration of the hypoglycemic episode.

Liver glycogen is the first substrate used to defend against hypoglycemia. Interestingly, hepatic glycogen levels in people with T1D are lower than those of non-T1D controls and their ability to mobilize liver glycogen to combat insulin-induced hypoglycemia is also diminished. Because of this, we carried out experiments in dogs to determine whether hepatic glycogen content is a determinant of the HGP response to insulin-induced hypoglycemia. Results of those studies showed that a 75% increase in liver glycogen (such as occurs in a non-T1D individual over the course of a day) generated a signal in the liver that was transmitted to the brain via afferent nerves which, in turn, led to an increase in the secretion of both epinephrine and glucagon. As expected, this increase in counterregulatory hormone secretion caused a 2.4-fold rise in HGP, despite insulin levels that were ~ 400 µU/mL at the liver.

The finding that an acute increase in hepatic glycogen can augment hypoglycemic counterregulation has important clinical implications. However, despite the potential of this therapeutic avenue to reduce the risk of iatrogenic hypoglycemia, it remains unclear at this point if such a strategy translates to humans with T1D. Therefore, the overarching theme of this proposal is to determine whether an acute increase in liver glycogen content can augment the hepatic and hormonal responses to insulin-induced hypoglycemia in humans with and without T1D. Herein we are proposing studies that will advance the field, with the specific aims being as follows:

Specific Aim #1: To determine the effect of increasing liver glycogen deposition on insulin-induced hypoglycemic counterregulation in humans with and without T1D.

The discovery of ways by which the risk of iatrogenic hypoglycemia can be reduced in people with T1D is a priority. The proposed experiments will improve our understanding of the mechanisms by which increased glycogen improves hypoglycemic counterregulation. If hypoglycemia is reduced by increased glycogen, it will focus attention on the ways in which liver glycogen levels can be normalized in people with T1D. This would be a significant step forward in the ongoing effort to reduce the risk of iatrogenic hypoglycemia in people with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race or ethnicity.
* Aged 21-40 years.
* Non-obese (BMI <28 kg/m2).

Exclusion Criteria:

* Pregnant women.
* Cigarette smoking.
* Taking inflammation-targeting steroids (e.g., prednisone).
* Taking medications targeting adrenergic signaling (e.g., beta-blockers, bronchodilators).
* Abnormal hematocrit or electrolyte levels.
* The presence of cardiovascular or peripheral vascular disease.
* The presence of neuropathy, retinopathy or nephropathy.
* Any metal in the body that would make magnetic resonance spectroscopy dangerous.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Epinephrine | 2 hours
  Hormone
Glucagon | 2 hours
  Hormone
Glucose Infusion Rate | 2 hours
  Whole-body responses

SECONDARY OUTCOMES:
Liver Glycogen | 2 hours
  Amount of sugar stored in the liver
Hepatic Glucose Production | 2 hours
  Amount of glucose released
Peripheral Glucose Uptake | 2 hours
  Amount of glucose being metabolized

CONTACTS AND LOCATIONS:
Overall Officials: Jason Winnick, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No